CLINICAL TRIAL: NCT02355847
Title: Cultural Competency, Risk Management, and Patient Safety Internet-Based Curriculum for OB/GYN Resident Physicians and Adverse Patient Events
Brief Title: Cultural Competency, Risk Management, and Patient Safety Internet-Based Curriculum for OB/GYN Resident Physicians
Acronym: PROM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brett Worly, MD (Other)
Responsible Party: Sponsor-Investigator, Brett Worly, MD, Primary Investigator, Ohio State University
Organization: Ohio State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 029701
Record Dates: First submitted 2014-11-18; First posted 2015-02-04 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-01

CONDITIONS: Risk Reduction
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthcare Worker Education (Other): Educational Lectures
  Interventions: Other: Lectures

INTERVENTIONS:
Other: Lectures — Lectures

SUMMARY:
Additional educational training lectures were provided to healthcare workers. Outcome measure of cultural competency was completed to assess patient safety, risk management, and cultural competency of healthcare providers in an urban academic Labor and Delivery Unit.

DETAILED DESCRIPTION:
Introduction: Patient safety, risk management, and cultural competency are essential topics for healthcare provider mastery in a high stakes, urban academic Labor and Delivery Unit.

Methods: A prospective cross sectional pilot study was performed with IRB exempt status to examine the effect of an internet based educational curriculum on topics including patient safety, risk management and cultural competency over 6 months amongst OB/GYN and Family Medicine medical students, nurses, and physicians. 76 healthcare providers participated. Assessments took place before and after curriculum implementation. Primary outcome measures were cultural competency as measured by the Tucker-Culturally Sensitive Health Care Inventory (TCSHCI) Provider Form, Pascal Metrics of Patient Safety survey for healthcare providers, patient satisfaction measured by the Press Ganey patient survey scores, and poor Labor and Delivery Outcomes. The curriculum intervention included five online lectures lasting 30-60 minutes pertaining to cultural competency, risk management, patient safety, and Team STEPPS training.

ELIGIBILITY:
Inclusion Criteria:. Inclusion criteria were OB/GYN medical students, Labor and Delivery nurses, and resident/ attending physicians in OB/GYN, Pediatrics, Anesthesia, and Family Medicine.

-

Exclusion Criteria:

* .Exclusion criteria were those providers that refused participation, or those that did not complete the course by June 2013.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Tucker-Culturally Sensitive Health Care Inventory (TCSHCI) Provider Form | 6 months
  Questionniare